CLINICAL TRIAL: NCT01795365
Title: Active Surveillance of 2 Groups of Patients With Localized Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Participants are no longer being examined and receiving intervention.
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Prof. Patrice Jichlinski, Chief of Urology Department, University of Lausanne Hospitals, Centre Hospitalier Universitaire Vaudois
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUV Active surveillance
Record Dates: First submitted 2013-01-23; First posted 2013-02-20 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Adenocarcinoma of the Prostate
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epstein + (group I) (Active Comparator): Epstein + (Group I) PSA <10 ng/ml; Gleason 3+3=6; Number of positive biopsies ≤3/12;
  % of tumor biopsy invasion <50% or ≤3mm; mp MRI negative; c-rTNM T1-T2a N0 M0
  Interventions: Other: Active surveillance
- Epstein - (group II) (Experimental): Epstein - (Group II) PSA <15 ng/ml; Gleason score max 3+4; Number of positive biopsies ≤5/12
  % of tumor biopsy invasion <50% and ≤8mm; mp MRI positive; T1-T2c N0 M0
  Interventions: Other: Active surveillance

INTERVENTIONS:
Other: Active surveillance

SUMMARY:
Active Surveillance manages selected men with prostate cancer expectantly with curative intent. This means men are carefully selected and subsequently actively observed in order to have the possibility to offer them curative treatment once the tumor seems to progress.

The goal of this study is to validate the treatment option Active Surveillance in men with localized, well differentiated prostate cancer, in order to limit the amount of overtreatment. A number of key points will be studied, such as the pathological findings in radical prostatectomy specimens, and the effect of expectancy on the quality of life.

DETAILED DESCRIPTION:
Objectives:

Primary

- To evaluate the equivalence of the time on active surveillance before an active treatment between group Epstein + and the expanded active surveillance group (Epstein -)

Secondary

* To evaluate the role of diffusion-weighted MRI (DW-MRI) in the initial diagnosis and the follow-up of patients under active surveillance
* To evaluate the role of BCAR-1 to predict the clinical outcome of localized prostate cancer
* To evaluate the proportion of patients who discontinued active surveillance
* To evaluate the mortality at 10, 15 and 20 years from the inclusion in the study
* To evaluate the time to radical treatment
* To evaluate the time to metastatic disease
* To evaluate patients quality of life

ELIGIBILITY:
Inclusion Criteria:

* Localized adenocarcinoma of the prostate with a Gleason score of 3+3 (group I patients) or 3+4 (group II patients)
* Percentage of tumor biopsy invasion <50% and/or with a size of maximum 8 mm
* With a number of positive tumor biopsies ≤3 (group I patients) or ≤ 5 (group II patients)
* TNM stage T1-2a N0 M0 (group I patients); TNM stage T1-2c N0 M0 (group II patients)
* PSA level at diagnosis < 10 ng/ml for group I patients; < 15 ng/ml for group II patients
* Tumor volume negative (group I patients); positive (group II patients)
* Absence of extra-capsular extension
* Life expectancy > 10 years
* Signed informed consent
* Patient has elected active surveillance as preferred management plan for the prostate cancer

Exclusion Criteria:

* Previous treatment for prostate cancer (including hormonal therapy, radiation therapy, surgery or chemotherapy)
* Patients with hypogonadism

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12; Primary Completion 2018-07 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
Proportion of patients on active surveillance in group Epstein + and Epstein - | 6 years

SECONDARY OUTCOMES:
Tumor volume increased, extra-capsular extension or presence of adenopathy assessed on DW-MRI | baseline, 12, 24, 48 months and every two years.
BCAR-1 test on biopsies | baseline, 12, 24 months and every 4 years
Percentage of patients who discontinued active surveillance by categories (patient's will, clinical or histological criterion) | Every 6 months for 6 years
Percentage of deceased patients 10, 15 and 20 years from the inclusion in the study in both groups | 10, 15, 20 years
Percentage of patients who progressed to a metastatic stage at different time points in both groups | Every year for 6 years
Quality of life assessment | Every 6 months for 6 years
  IPSS score/IIEF-5 score( QLQ-C30 + PR25)

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Jichlinski, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Switzerland